CLINICAL TRIAL: NCT06856122
Title: Pharmacogenomics to Improve Supportive Care Symptoms. A Prospective Observational Study
Brief Title: Pharmacogenomics to Improve Supportive Care Symptoms.
Acronym: PISCES
Status: Enrolling by invitation | Type: Observational
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: Manchester Centre for Genomic Medicine - St. Mary's Hospital University of Manchester (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024GRANT089
Record Dates: First submitted 2025-02-05; First posted 2025-03-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-02

CONDITIONS: Palliative Care; Supportive Care
Keywords: Pharmacogenomics; pharmacogenetics; palliative; supportive care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study participants: Patients with serious and/or life limiting condition conditions, such as incurable cancer undergoing palliative or supportive care treatment. They will have a 5mL blood sample collected.

SUMMARY:
To understand the clinical utility of multi-gene pharmacogenetic testing in patients receiving palliative and supportive care across palliative care settings (inpatient hospital, outpatient), specifically to calculate a drug-gene interaction ratio, based on extant prescriptions paired with an individual's pharmacogenetic results.

DETAILED DESCRIPTION:
This is a prospective, observational cross-sectional study of patients with serious and/or life limiting condition conditions, such as incurable cancer undergoing palliative or supportive care treatment at a University Teaching Hospital in England, UK. Participants will be recruited at point of referral to in-patient or outpatient palliative care services (i.e. at point of presentation with symptom control issues).

All participant study activities:

All participants will undergo testing of a panel of genetic variants relevant to drugs used in symptom control (see https://cpicpgx.org/genes-drugs/ ). This will involve collecting a 5mL blood sample (the intervention) from individuals. All participants will be consented to examination of their records within local hospitals and/or primary care to extract study relevant data (described below).

The start of follow-up will be from the date of the blood sample (the intervention). Standard demographic information including ethnicity will be collected at baseline.

Participation in study will be for the duration of being under palliative care treatment, up to a maximum of 90days from recruitment date.

All participant sample will be stored and genetic analysis will take place after the end of recruitment and health data collection.

The study team will then calculate a drug-gene interaction ratio (DGI) (i.e. The total number of genetic variation results that pair with a relevant prescribed medication for that same individual, divided by total number of individuals tested).

ELIGIBILITY:
Inclusion Criteria: Aged 18 or older; incurable, life limiting condition, clinical care provided at NNUH.

Exclusion Criteria: Lacking capacity to consent to research (unless there is an appropriate consultee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be from Norfolk and Norwich University Hospitals NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Drug-gene interaction ratio (DGI) | This will be calculated for all current medications prescribed at the point of recruitment.
  The total number of genetic variation results that pair with a relevant prescribed medication for that same individual, divided by total number of individuals tested.

SECONDARY OUTCOMES:
Frequency of changes in prescription medication that are potentially affected by drug-gene interaction | from enrolment until 90 days post blood test
  Number of participants who have a change in prescribed medication (dose or formulation) during 90 day follow up period that could be theoretically paired to possession of a clinically relevant drug-gene interaction

CONTACTS AND LOCATIONS:
Overall Officials: Dr Martyn Patel, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK); Dr Caroline Barry, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (2):
- United Kingdom (2):
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - The Manchester Centre for Genomic Medicine, Manchester

REFERENCES:
- [Background] Barry C, Patel M. Pharmacogenomics and symptom management in palliative and supportive care: A scoping review. BMJ Support Palliat Care. 2025 Feb 26;15(2):158-167. doi: 10.1136/spcare-2024-005205. PMID 39805678